CLINICAL TRIAL: NCT06736327
Title: A Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of SKB500 for Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study on the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of SKB500 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB500-Ⅰ-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB500 (Experimental): Subjects will receive SKB500 once every three weeks (Q3W).
  Interventions: Drug: SKB500

INTERVENTIONS:
Drug: SKB500 — The administration route of SKB500 is intravenous infusion, with a dosing frequency of Q3W.

SUMMARY:
This study aims to evaluate the safety, tolerability, PK profile, immunogenicity, and antitumor activity of SKB500 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open-label Phase I clinical trial to evaluate the safety, tolerability, PK profile, immunogenicity, and antitumor activity of SKB500 in subjects with advanced solid tumors. The study includes a dose-escalation phase, a dose-expansion phase, and an indication-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 75 years old.
2. Histologically or cytologically confirmed advanced solid tumors for which standard treatment either does not exist or has proven ineffective or intolerable.
3. Subjects should ideally provide a tumor tissue sample for biomarker testing during the screening period.
4. Has at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
5. ECOG performance status score of 0 or 1.
6. Expected survival of at least 12 weeks.
7. Has adequate hematopoietic, renal and hepatic functions.
8. Have recovered to grade ≤ 1 of prior anti-cancer treatment toxicities.
9. Male and female subjects must agree to use highly effective contraceptive methods throughout the study.
10. Subjects must voluntarily enter the study, sign the informed consent form, and be able to comply with the visits and procedures.

Exclusion Criteria:

1. Subjects with known active CNS metastases, carcinomatous meningitis, leptomeningeal metastases, or spinal cord compression.
2. Subjects with other malignancies within 5 years before the first dose.
3. Any severe and/or uncontrolled concurrent disease that may interfere with the subject's participation in the study.
4. Active hepatitis B, or hepatitis C; active tuberculosis, or human immunodeficiency virus (HIV) test positive, or known acquired immunodeficiency syndrome (AIDS).
5. History of allergy to any component of SKB500 or history of severe hypersensitivity reactions to other monoclonal antibodies.
6. Subjects with a history of interstitial lung disease, non-infectious pneumonia, or other pulmonary diseases significantly affecting lung function.
7. History of allogeneic organ transplantation or hematopoietic stem cell transplantation.
8. Uncontrolled pleural effusion, ascites, or pericardial effusion.
9. Have received ADCs with the same target or the same toxins.
10. Have received chemotherapy, small molecule targeted therapy, and traditional Chinese medicine preparations within 14 days or 5 half-lives before the first dose; have received any immunotherapy, large molecule anticancer drug treatment, or more than 30% bone marrow radiation or extensive radiotherapy within 28 days before the first dose.
11. Have undergone major surgery or severe trauma within 28 days before the first dose.
12. Have received other clinical trial medications within 28 days before the first dose.
13. Has previously received anti-cancer or live vaccines within 28 days before the first dose
14. Have received systemic steroids or other immunosuppressive treatments within 14 days before the first dose.
15. Have received potent CYP3A4 inhibitors, inducers, or BCRP inhibitors within 14 days or 5 half-lives before the first dose.
16. Pregnant or lactating female.
17. Any disease or condition that, in the investigator's opinion, would compromise subject safety or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of adverse events (AEs) | Up to 3 years
Evaluate the incidence of serious adverse events (SAEs) | Up to 3 years
Evaluate the incidence of treatment related adverse events (TRAEs) | Up to 3 years
Evaluate the incidence of dose-limiting toxicities (DLTs) | Day 1 to Day 21 in Cycle 1 in the dose escalation part

SECONDARY OUTCOMES:
Investigate the antitumor activity of SKB500 | Up to 3 years
To evaluate the Tmax of SKB500 | Up to 3 years
To evaluate the Cmax of SKB500 | Up to 3 years
To evaluate the Cmin of SKB500 | Up to 3 years
To evaluate the AUC of SKB500 | Up to 3 years
To evaluate the t1/2 of SKB500 | Up to 3 years
To evaluate the CL of SKB500 | Up to 3 years
To evaluate the Vz of SKB500 | Up to 3 years
To evaluate the ADA of SKB500 | Up to 3 years

OTHER OUTCOMES:
To evaluate the relationship between the biomarker and the antitumor activity | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- JILIN Cancer Hospital, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided